CLINICAL TRIAL: NCT03249792
Title: A Phase 1 Open-label, Multicenter Study of MK-2118 Administered by Intratumoral Injection as Monotherapy and in Combination With Pembrolizumab or by Subcutaneous Injection in Combination With Pembrolizumab for Patients With Advanced/Metastatic Solid Tumors or Lymphomas
Brief Title: Study of MK-2118 Administered as Intratumoral Injection as Monotherapy and in Combination With Pembrolizumab (MK-3475) or by Subcutaneous Injection in Combination With Pembrolizumab in the Treatment of Adults With Advanced/Metastatic Solid Tumors or Lymphomas (MK-2118-001)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2118-001; MK-2118-001 (Other: Merck)
Record Dates: First submitted 2017-08-09; First posted 2017-08-15 (Actual); Results first posted 2024-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (25):
- Arm 1 MK-2118 100 µg Intra-tumoral (IT) Monotherapy (Experimental): Participants receive MK-2118 100 µg via IT injection once weekly (Q1W) on Days 1, 8 and 15 of Cycles 1-3 followed by once every 3 weeks (Q3W) on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT)
- Arm 1 MK-2118 300 µg IT Monotherapy (Experimental): Participants receive MK-2118 300 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT)
- Arm 1 MK-2118 900 µg IT Monotherapy (Experimental): Participants receive MK-2118 900 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT)
- Arm 1 MK-2118 2700 µg IT Monotherapy (Experimental): Participants receive MK-2118 2700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT)
- Arm 1 MK-2118 5400 µg IT Monotherapy (Experimental): Participants receive MK-2118 5400 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT)
- Arm 1 MK-2118 7700 µg IT Monotherapy (Experimental): Participants receive MK-2118 7700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT)
- Arm 1 MK-2118 10000 µg IT Monotherapy (Experimental): Participants receive MK-2118 10000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT)
- Arm 1 MK-2118 15000 µg IT Monotherapy (Experimental): Participants receive MK-2118 15000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT)
- Arm 1 MK-2118 20000 µg IT Monotherapy (Experimental): Participants receive MK-2118 20000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT)
- Arm 2 MK-2118 2700 µg IT + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 2700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT); Biological: Pembrolizumab
- Arm 2 MK-2118 5400 µg IT + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 5400 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT); Biological: Pembrolizumab
- Arm 2 MK-2118 7700 µg IT + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 7700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT); Biological: Pembrolizumab
- Arm 2 MK-2118 10000 µg IT + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 10000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT); Biological: Pembrolizumab
- Arm 2 MK-2118 15000 µg IT + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 15000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT); Biological: Pembrolizumab
- (Not Enrolled) Arm 3 MK-2118 Visceral IT + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-2 followed by Q3W on Day 1 of Cycle 3 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
  Interventions: Drug: MK-2118 (IT); Biological: Pembrolizumab
- Arm 4: MK-2118 5000 µg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 5000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed Q3W Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
  Interventions: Drug: MK-2118 (SC); Biological: Pembrolizumab
- Arm 4: MK-2118 10000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 10000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed Q3W Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
  Interventions: Drug: MK-2118 (SC); Biological: Pembrolizumab
- Arm 4: MK-2118 15000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 15000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed Q3W Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
  Interventions: Drug: MK-2118 (SC); Biological: Pembrolizumab
- Arm 4: MK-2118 20000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 20000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed Q3W Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
  Interventions: Drug: MK-2118 (SC); Biological: Pembrolizumab
- Arm 4: MK-2118 30000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 30000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed Q3W Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
  Interventions: Drug: MK-2118 (SC); Biological: Pembrolizumab
- Arm 4: MK-2118 45000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 45000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed Q3W Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
  Interventions: Drug: MK-2118 (SC); Biological: Pembrolizumab
- Arm 4: MK-2118 60000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 60000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed Q3W Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
  Interventions: Drug: MK-2118 (SC); Biological: Pembrolizumab
- Arm 4: MK-2118 90000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 90000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed Q3W Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
  Interventions: Drug: MK-2118 (SC); Biological: Pembrolizumab
- Arm 4: MK-2118 120000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 120000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed Q3W Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
  Interventions: Drug: MK-2118 (SC); Biological: Pembrolizumab
- Arm 4: MK-2118 150000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (Experimental): Participants receive MK-2118 150000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed Q3W Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and receive pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
  Interventions: Drug: MK-2118 (SC); Biological: Pembrolizumab

INTERVENTIONS:
Drug: MK-2118 (IT) — IT injection
  Arms: (Not Enrolled) Arm 3 MK-2118 Visceral IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 1 MK-2118 100 µg Intra-tumoral (IT) Monotherapy; Arm 1 MK-2118 10000 µg IT Monotherapy; Arm 1 MK-2118 15000 µg IT Monotherapy; Arm 1 MK-2118 20000 µg IT Monotherapy; Arm 1 MK-2118 2700 µg IT Monotherapy; Arm 1 MK-2118 300 µg IT Monotherapy; Arm 1 MK-2118 5400 µg IT Monotherapy; Arm 1 MK-2118 7700 µg IT Monotherapy; Arm 1 MK-2118 900 µg IT Monotherapy; Arm 2 MK-2118 10000 µg IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 2 MK-2118 15000 µg IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 2 MK-2118 2700 µg IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 2 MK-2118 5400 µg IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 2 MK-2118 7700 µg IT + Pembrolizumab 200 mg IV Combination Therapy
Drug: MK-2118 (SC) — SC injection
  Arms: Arm 4: MK-2118 10000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 120000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 15000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 150000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 20000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 30000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 45000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 5000 µg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 60000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 90000 µg SC + Pembrolizumab 200 mg IV Combination Therapy
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475
  Arms: (Not Enrolled) Arm 3 MK-2118 Visceral IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 2 MK-2118 10000 µg IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 2 MK-2118 15000 µg IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 2 MK-2118 2700 µg IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 2 MK-2118 5400 µg IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 2 MK-2118 7700 µg IT + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 10000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 120000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 15000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 150000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 20000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 30000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 45000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 5000 µg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 60000 µg SC + Pembrolizumab 200 mg IV Combination Therapy; Arm 4: MK-2118 90000 µg SC + Pembrolizumab 200 mg IV Combination Therapy

SUMMARY:
The purposes of this study are to: 1) assess the safety and tolerability and 2) establish a preliminary recommended Phase 2 dose (RP2D) and/or a maximum tolerated dose (MTD) or a maximum administered dose (MAD) of MK-2118 when administered via intratumoral (IT) injection as monotherapy and in combination with pembrolizumab (MK-3475) intravenous (IV) infusion, or via subcutaneous (SC) injection in combination with pembrolizumab IV infusion in the treatment of adult participants with advanced/metastatic solid tumors or lymphomas.

Participants will receive either MK-2118 monotherapy or MK-2118 in combination with pembrolizumab for up to 35 cycles for Arms 1-3 or up to 36 cycles for Arm 4 (up to approximately 2 years).

All participants will undergo at least a 24-hour observation period following the first three administrations of MK-2118 (Arms 1-3: Cycle 1 Days 1, 8, and 15. Arm 4: Cycle 1 Days 1 and 8; and Cycle 2 Day 1).

Qualified participants who experience radiographic or clinical progression in Arm 1 (MK-2118 Intra-tumoral [IT] monotherapy) may switch over to Arm 2 (MK-2118 IT + Pembrolizumab IV Combination Therapy) at an eligible dose.

Pharmacokinetic (PK) outcome measures will not be analyzed separately for the switch-over treatment arms, per protocol.

DETAILED DESCRIPTION:
Arm 3 did not enroll any participants.

Data for the pembrolizumab Cmin outcome measure were not collected.

ELIGIBILITY:
Inclusion Criteria:

Arms 1 and 2 Participants:

* Has any histologically or cytologically confirmed advanced/metastatic solid tumor by pathology report and has received, or have been intolerant to all treatment known to confer clinical benefit. Solid tumors and lymphomas of any type are eligible for enrollment. For cutaneous T-cell lymphoma (CTCL), histopathological diagnosis should be confirmed in a skin biopsy representative of disease.
* Has Stage III or Stage IV disease that is not surgically resectable. Stage IIB (T3N0M0B0-1) CTCL participants are eligible.

Arm 3 Participants:

- Has metastatic liver and/or liver lesion involvement that does not exceed one third of the total liver volume in participants to be treated by liver IT injection. Hepatocellular carcinoma participants are excluded from eligibility of IT liver injection.

All Participants:

* Has Stage III or Stage IV disease that is not surgically resectable.
* Has ≥1 injectable lesion that is amenable to injection and biopsy via visual inspection for a cutaneous lesion, or via ultrasound guidance for a subcutaneous lesion.
* Has ≥1 discrete, distant noninjected lesion that is amenable to biopsy via visual inspection or amenable to biopsy via image guidance.
* Has Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Demonstrates adequate organ function.
* A male participant is eligible to participate if he agrees to the following during the intervention period and for at least 120 days after the last dose of study intervetnion:

  1. Refrain from donating sperm.
  2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle and agree to remain abstinent OR must agree to use contraception unless confirmed to be azoospermic.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  1. Is not a woman of childbearing potential (WOCBP).
  2. Is a WOCBP and using a contraceptive method that is highly effective with low user dependency, or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis), during the intervention period and for at least 120 days after the last dose of study intervention, AND agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period.
* Human Immunodeficiency Virus (HIV)-infected participants must meet these additional criteria:

  1. Has HIV-1 infection documented by laboratory test.
  2. Has well-controlled HIV on antiretroviral therapy (ART), defined as: 1) must have a CD4+ T-cell count >350 cells/mm^3 at time of screening; 2) must have achieved and maintained virologic suppression defined as confirmed HIV ribonucleic acid (RNA) level <50 or below the lower limit of quantification (LLOQ) using the locally available assay at the time of screening and for ≥12 weeks prior to screening; and 3) must have been on a stable regimen, without changes in drugs or dose modification, for ≥4 weeks prior to study entry (Day 1).

Exclusion Criteria:

* Has history of a second malignancy, unless potentially curative treatment has been completed, with no evidence of malignancy for 2 years (except for successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, or in situ cervical cancer).
* Has clinically active central nervous system metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity reaction to treatment with a monoclonal antibody (mAb).
* Has active autoimmune disease that has required systemic treatment in the past 2 years.
* Has history of vasculitis.
* Has active infection requiring therapy.
* Has history of (noninfectious) pneumonitis that required steroids or current pneumonitis.
* Has undergone prior allogeneic hematopoietic stem cell transplantation within the last 5 years.
* Has known Hepatitis B or C infection.
* Has known psychiatric or substance abuse disorders that would interfere in cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study.
* Is not fully recovered from any effects of major surgery, and is free of significant detectable infection.
* HIV-infected participants with history of Kaposi's sarcoma and/or multicentric Castleman's disease.
* HIV-infected participants who have had an HIV-related opportunistic infection within 6 months.
* Has had chemotherapy, definitive radiation, or biological cancer therapy within 4 weeks (2 weeks for palliative radiation) prior to the first dose of study treatment, or has not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 from the AEs due to cancer therapeutics administered >4 weeks earlier.
* Has been treated within 2 weeks of Cycle 1 Day1 with any of the following: strong/moderate Cytochrome P450 2C9 (CYP2C9) inhibitors, such as: amiodarone, felbamate, fluconazole, miconazole, piperine, oxandrolone, fluorouracil and its derivatives (combination drug tegafur/gimeracil/oteracil [TS-1], Uftoral [UFT], tegafur, carmofur, doxifluridine, capecitabine), sulfaphenazole, cyclosporine, bucurol, tienilic acid; UGT1A3 inhibitors (including ritonavir, quinidine, probenecid, and valproic acid); or strong carbonyl reductase (CBR) inhibitors (including quercetin, menadione, glycyrrhetinic acid, and flufenamic acid).
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and has received study therapy or has used an investigational device within 28 days of administration of MK-2118.
* Is expected to require any other form of antineoplastic therapy while on study.
* Is on chronic systemic steroid therapy in excess of replacement doses (prednisone ≤10 mg/day is acceptable), or on any other form of immunosuppressive medication. For CTCL, continued use of either prednisone ≤10 mg/day or continued use of topical steroids is acceptable.
* Has received a live vaccine within 28 days prior to first dose.
* Has been treated with a stimulator of interferon genes (STING) agonist (eg, MK-1454, ADU-S100 [synthetic cyclic dinucleotide (CDN)]).
* Has a history of re-irradiation for head and neck squamous cell carcinoma (HNSCC) at the projected injection site.
* Has a tumor(s) in direct contact or encases a major blood vessel and has ulceration and/or fungation onto the skin surface at the projected injection site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (8):
- United States (7):
  - University of California San Diego Moores Cancer Center ( Site 0004), La Jolla, California
  - UCLA ( Site 0003), Los Angeles, California
  - University of Chicago ( Site 0002), Chicago, Illinois
  - New York Presbyterian Hospital/Columbia University ( Site 0001), New York, New York
  - UPMC Hillman Cancer Centers ( Site 0007), Pittsburgh, Pennsylvania
  - Mary Crowley Cancer Research Center ( Site 0005), Dallas, Texas
  - MD Anderson Cancer Centr. ( Site 0006), Houston, Texas
- Sheba Medical Center ( Site 0301), Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Luke JJ, Sweis RF, Hecht JR, Schneider R, Stein MN, Golan T, Yap TA, Khilnani A, Huang M, Zhao R, Jemielita T, Patel SP. Intratumoral or Subcutaneous MK-2118, a Noncyclic Dinucleotide STING Agonist, with or without Pembrolizumab, for Advanced or Metastatic Solid Tumors or Lymphomas. Clin Cancer Res. 2025 Apr 1;31(7):1233-1242. doi: 10.1158/1078-0432.CCR-24-2824. PMID 39846804
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Arm 3 did not enroll any participants.
  Per protocol, pharmacokinetic (PK) outcome measures were not analyzed separately for the switch-over treatment arms.
Groups:
- Arm 1 MK-2118 100 µg Intra-tumoral (IT) Monotherapy: Participants received MK-2118 100 µg via IT injection once weekly (Q1W) on Days 1, 8 and 15 of Cycles 1-3 followed by once every 3 weeks (Q3W) on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 300 µg IT Monotherapy: Participants received MK-2118 300 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 900 µg IT Monotherapy: Participants received MK-2118 900 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 2700 µg IT Monotherapy: Participants received MK-2118 2700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 5400 µg IT Monotherapy: Participants received MK-2118 5400 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 7700 µg IT Monotherapy: Participants received MK-2118 7700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 10000 µg IT Monotherapy: Participants received MK-2118 10000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 15000 µg IT Monotherapy: Participants received MK-2118 15000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 20000 µg IT Monotherapy: Participants received MK-2118 20000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 2 MK-2118 2700 µg IT + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 2700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 2 MK-2118 5400 µg IT + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 5400 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 2 MK-2118 7700 µg IT + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 7700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 2 MK-2118 10000 µg IT + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 10000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 2 MK-2118 15000 µg IT + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 15000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- (Not Enrolled) Arm 3 MK-2118 Visceral IT + Pembrolizumab 200 mg IV Combination Therapy: Participants were to receive MK-2118 via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-2 followed by Q3W on Day 1 of Cycle 3 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 4: MK-2118 5000 µg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 5000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 10000 µg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 10000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 15000 µg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 15000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 20000 µg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 20000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 30000 µg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 30000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 45000 µg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 45000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 60000 µg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 60000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 90000 µg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 90000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 120000 µg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 120000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 150000 µg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 150000 µg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Switch-over Arm 1 MK-2118 300 µg IT To Arm 2 900 µg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK-2118 300 µg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 900 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 2700 µg IT To Arm 2 2700 µg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK-2118 2700 µg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 2700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 5400 µg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK-2118 15000 µg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 5400 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 900 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK-2118 900 µg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 7700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 7700 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK-2118 7700 µg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 7700 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK-2118 15000 µg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 10000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK-2118 20000 µg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 10000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 15000 µg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK-2118 20000 µg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 15000 µg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
Period: Arms 1, 2, and 4
Arm/Group | Arm 1 MK-2118 100 µg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 µg IT Monotherapy | Arm 1 MK-2118 900 µg IT Monotherapy | Arm 1 MK-2118 2700 µg IT Monotherapy | Arm 1 MK-2118 5400 µg IT Monotherapy | Arm 1 MK-2118 7700 µg IT Monotherapy | Arm 1 MK-2118 10000 µg IT Monotherapy | Arm 1 MK-2118 15000 µg IT Monotherapy | Arm 1 MK-2118 20000 µg IT Monotherapy | Arm 2 MK-2118 2700 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 µg IT + Pembrolizumab 200 mg IV Combination Therapy | (Not Enrolled) Arm 3 MK-2118 Visceral IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 µg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Switch-over Arm 1 MK-2118 300 µg IT To Arm 2 900 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 2700 µg IT To Arm 2 2700 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 5400 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 900 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 7700 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 15000 µg IT + Pembrolizumab 200 mg IV
Started | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 18 | 13 | 0 | 4 | 8 | 14 | 7 | 6 | 3 | 3 | 3 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 16 | 13 | 0 | 4 | 8 | 14 | 7 | 6 | 3 | 3 | 3 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 18 | 13 | 0 | 4 | 8 | 14 | 7 | 6 | 3 | 3 | 3 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 2 | 3 | 2 | 2 | 4 | 2 | 1 | 7 | 7 | 12 | 7 | 0 | 4 | 4 | 12 | 6 | 4 | 2 | 3 | 1 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 0 | 2 | 1 | 4 | 3 | 5 | 3 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Switch Over Period
Arm/Group | Arm 1 MK-2118 100 µg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 µg IT Monotherapy | Arm 1 MK-2118 900 µg IT Monotherapy | Arm 1 MK-2118 2700 µg IT Monotherapy | Arm 1 MK-2118 5400 µg IT Monotherapy | Arm 1 MK-2118 7700 µg IT Monotherapy | Arm 1 MK-2118 10000 µg IT Monotherapy | Arm 1 MK-2118 15000 µg IT Monotherapy | Arm 1 MK-2118 20000 µg IT Monotherapy | Arm 2 MK-2118 2700 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 µg IT + Pembrolizumab 200 mg IV Combination Therapy | (Not Enrolled) Arm 3 MK-2118 Visceral IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 µg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Switch-over Arm 1 MK-2118 300 µg IT To Arm 2 900 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 2700 µg IT To Arm 2 2700 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 5400 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 900 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 7700 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 15000 µg IT + Pembrolizumab 200 mg IV
Started (The protocol-specified optional switch over period included qualified participants from Arm 1 who switched over to receive combination therapy in Arm 2 at an eligible dose.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analyzed in all participants allocated to Arms 1, 2, and 4. Arm 3 did not enroll any participants. Per protocol, baseline characteristics were not analyzed separately for the switch over period.
Groups:
- Arm 1 MK-2118 100 μg Intra-tumoral (IT) Monotherapy: Participants received MK-2118 100 μg via IT injection once weekly (Q1W) on Days 1, 8 and 15 of Cycles 1-3 followed by once every 3 weeks (Q3W) on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 300 μg IT Monotherapy: Participants received MK-2118 300 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 900 μg IT Monotherapy: Participants received MK-2118 900 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 2700 μg IT Monotherapy: Participants received MK-2118 2700 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 5400 μg IT Monotherapy: Participants received MK-2118 5400 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 7700 μg IT Monotherapy: Participants received MK-2118 7700 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 10000 μg IT Monotherapy: Participants received MK-2118 10000 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 15000 μg IT Monotherapy: Participants received MK-2118 15000 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 1 MK-2118 20000 μg IT Monotherapy: Participants received MK-2118 20000 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 2 MK-2118 2700 μg IT + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 2700 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 2 MK-2118 5400 μg IT + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 5400 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 2 MK-2118 7700 μg IT + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 7700 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 2 MK-2118 10000 μg IT + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 10000 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 2 MK-2118 15000 μg IT + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 15000 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for a total of up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Arm 4: MK-2118 5000 μg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 5000 μg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 10000 μg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 10000 μg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 15000 μg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 15000 μg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 20000 μg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 20000 μg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 30000 μg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 30000 μg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 45000 μg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 45000 μg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 60000 μg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 60000 μg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 90000 μg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 90000 μg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 120000 μg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 120000 μg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Arm 4: MK-2118 150000 μg SC + Pembrolizumab 200 mg IV Combination Therapy: Participants received MK-2118 150000 μg via SC injection Q1W on Days 1 and 8 of Cycle 1 followed by Q1W on Days 1, 8 and 15 of Cycles 2-4, followed by Q3W on Day 1 of Cycle 5 and beyond, for a total of up to 36 cycles (up to ~2 years) and received pembrolizumab 200 mg via IV infusion on Day 1 of Cycle 2 and beyond for a total of up to 36 cycles (up to ~2 years). Cycle 1 is 2 weeks long and Cycles 2 to 36 are 3 weeks long.
- Total: Total of all reporting groups
Arm/Group | Arm 1 MK-2118 100 μg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 μg IT Monotherapy | Arm 1 MK-2118 900 μg IT Monotherapy | Arm 1 MK-2118 2700 μg IT Monotherapy | Arm 1 MK-2118 5400 μg IT Monotherapy | Arm 1 MK-2118 7700 μg IT Monotherapy | Arm 1 MK-2118 10000 μg IT Monotherapy | Arm 1 MK-2118 15000 μg IT Monotherapy | Arm 1 MK-2118 20000 μg IT Monotherapy | Arm 2 MK-2118 2700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 μg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Total
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 18 | 13 | 4 | 8 | 14 | 7 | 6 | 3 | 3 | 3 | 4 | 4 | 140
Age, Customized [Count of Participants; unit: Participants]
  0 to 17 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18 to 64 years | 1 | 0 | 1 | 2 | 2 | 2 | 4 | 2 | 4 | 2 | 9 | 7 | 9 | 10 | 3 | 4 | 13 | 6 | 4 | 1 | 2 | 2 | 2 | 1 | 93
  65 to 84 years | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 0 | 4 | 4 | 8 | 3 | 1 | 4 | 1 | 0 | 2 | 2 | 0 | 1 | 2 | 3 | 44
  85 years and over | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 2 | 0 | 3 | 3 | 1 | 2 | 1 | 7 | 4 | 11 | 7 | 1 | 4 | 5 | 0 | 1 | 0 | 1 | 1 | 3 | 3 | 61
  Male | 1 | 0 | 1 | 0 | 3 | 0 | 3 | 3 | 4 | 1 | 6 | 7 | 7 | 6 | 3 | 4 | 9 | 7 | 5 | 3 | 2 | 2 | 1 | 1 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Participants are indicated as "not reported" due to the risk of identification of a person.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 18 | 13 | 4 | 8 | 14 | 7 | 6 | 3 | 3 | 3 | 4 | 4 | 140
Race (NIH/OMB) [Count of Participants; unit: Participants] — Participants are indicated as "not reported" due to the risk of identification of a person.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 18 | 13 | 4 | 8 | 14 | 7 | 6 | 3 | 3 | 3 | 4 | 4 | 140

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience One or More Dose-limiting Toxicities (DLTs)
Description: A DLT is defined as the following toxicities, if related to study treatment: Grade 4 nonhematologic toxicity; Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia (Grade 4 thrombocytopenia, Grade 3 thrombocytopenia with significant bleeding); non-hematologic adverse event (AE) ≥Grade 3 (with exceptions); Grade 3 or Grade 4 nonhematologic abnormality; febrile neutropenia Grade 3 or 4; any toxicity causing treatment discontinuation or missing ≥1 dose; any toxicity causing a >2 week delay initiating pembrolizumab; any elevated aspartate aminotransferase or alanine aminotransferase value that is ≥3× upper limit of normal (ULN) and an elevated total bilirubin value that is ≥2× ULN & an alkaline phosphatase value that is <2× ULN with no alternative explanation; any ≥Grade 2 immune-mediated uveitis; Grade 5 toxicity. Per protocol, DLTs were analyzed separately for the switch-over treatment arms. The number of participants who experienced one or more DLTs is reported.
Time Frame: Up to ~35 days
Population: All allocated participants who received ≥1 dose of study treatment, who were observed for DLTs for up to 35 days after the first dose of assigned treatment, and had data available for this outcome. Per protocol, DLTs were analyzed separately for the switch-over treatment arms.
Measure: Count of Participants; unit: Participants
Groups:
- Switch-over Arm 1 MK-2118 300 μg IT To Arm 2 900 μg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK 2118 300 μg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 900 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 2700 μg IT To Arm 2 2700 μg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK 2118 2700 μg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 2700 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 5400 μg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK 2118 15000 μg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 5400 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 900 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK 2118 900 μg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 7700 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 7700 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK 2118 7700 μg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 7700 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK 2118 15000 μg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 10000 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK 2118 20000 μg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 10000 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
- Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 15000 μg IT + Pembrolizumab 200 mg IV: Qualified participants who received MK 2118 20000 μg via IT injection in Arm 1 but experienced disease progression switched over to Arm 2 and received combination therapy of MK-2118 15000 μg via IT injection Q1W on Days 1, 8 and 15 of Cycles 1-3 followed by Q3W on Day 1 of Cycle 4 and beyond, for a total of up to ~35 cycles (up to ~2 years) and pembrolizumab 200 mg via IV infusion on Day 1 of each cycle for up to ~35 cycles (up to ~2 years). Each cycle is 3 weeks long.
Arm/Group | Arm 1 MK-2118 100 μg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 μg IT Monotherapy | Arm 1 MK-2118 900 μg IT Monotherapy | Arm 1 MK-2118 2700 μg IT Monotherapy | Arm 1 MK-2118 5400 μg IT Monotherapy | Arm 1 MK-2118 7700 μg IT Monotherapy | Arm 1 MK-2118 10000 μg IT Monotherapy | Arm 1 MK-2118 15000 μg IT Monotherapy | Arm 1 MK-2118 20000 μg IT Monotherapy | Arm 2 MK-2118 2700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 μg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Switch-over Arm 1 MK-2118 300 μg IT To Arm 2 900 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 2700 μg IT To Arm 2 2700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 5400 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 900 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 7700 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 15000 μg IT + Pembrolizumab 200 mg IV
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 15 | 13 | 3 | 8 | 13 | 7 | 6 | 3 | 3 | 3 | 3 | 3 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

2. Primary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Per protocol, safety was analyzed separately for the switch-over treatment arms. The number of participants who experienced one or more AEs is reported.
Time Frame: Up to ~65 months
Population: All allocated participants who received ≥1 dose of study treatment. Per protocol, safety was analyzed separately for the switch-over treatment arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 MK-2118 100 μg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 μg IT Monotherapy | Arm 1 MK-2118 900 μg IT Monotherapy | Arm 1 MK-2118 2700 μg IT Monotherapy | Arm 1 MK-2118 5400 μg IT Monotherapy | Arm 1 MK-2118 7700 μg IT Monotherapy | Arm 1 MK-2118 10000 μg IT Monotherapy | Arm 1 MK-2118 15000 μg IT Monotherapy | Arm 1 MK-2118 20000 μg IT Monotherapy | Arm 2 MK-2118 2700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 μg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Switch-over Arm 1 MK-2118 300 μg IT To Arm 2 900 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 2700 μg IT To Arm 2 2700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 5400 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 900 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 7700 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 15000 μg IT + Pembrolizumab 200 mg IV
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 16 | 13 | 4 | 8 | 14 | 7 | 6 | 3 | 3 | 3 | 4 | 4 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Participants | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 16 | 12 | 4 | 8 | 14 | 7 | 6 | 3 | 3 | 3 | 4 | 4 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 1

3. Primary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Per protocol, tolerability was analyzed separately for the switch-over treatment arms. The number of participants who discontinued study treatment due to an AE is reported.
Time Frame: Up to ~27 months
Population: All allocated participants who received ≥1 dose of study treatment. Per protocol, tolerability was analyzed separately for the switch-over treatment arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 MK-2118 100 μg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 μg IT Monotherapy | Arm 1 MK-2118 900 μg IT Monotherapy | Arm 1 MK-2118 2700 μg IT Monotherapy | Arm 1 MK-2118 5400 μg IT Monotherapy | Arm 1 MK-2118 7700 μg IT Monotherapy | Arm 1 MK-2118 10000 μg IT Monotherapy | Arm 1 MK-2118 15000 μg IT Monotherapy | Arm 1 MK-2118 20000 μg IT Monotherapy | Arm 2 MK-2118 2700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 μg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Switch-over Arm 1 MK-2118 300 μg IT To Arm 2 900 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 2700 μg IT To Arm 2 2700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 5400 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 900 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 7700 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 15000 μg IT + Pembrolizumab 200 mg IV
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 16 | 13 | 4 | 8 | 14 | 7 | 6 | 3 | 3 | 3 | 4 | 4 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: MK-2118 Minimum Plasma Concentration (Cmin)
Description: Cmin of MK-2118 was defined as the minimum concentration of MK-2118 observed in plasma. Blood samples were collected pre-dose and at specified timepoints post dose for estimation of MK-2118 Cmin. Per protocol, PK outcomes were not analyzed separately for the switch-over treatment arms.
Time Frame: Cycle 1 Day 1: Predose, 0.5, 1, 2, 4, 6, 8, 12, 24 hours postdose; Cycle 2 Day 1, Cycle 3 Day 1: Predose, 0.5, 1, 2, 4, 6, 8 hours postdose (Arms 1 and 2: length of Cycle= 3 weeks, Arm 4: length of Cycle 1= 2 weeks, length of Cycles 2 and 3= 3 weeks)
Population: The subset of participants who complied with the protocol and had MK-2118 Cmin data available. Per protocol, PK outcomes were not analyzed separately for the switch-over treatment arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 MK-2118 100 μg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 μg IT Monotherapy | Arm 1 MK-2118 900 μg IT Monotherapy | Arm 1 MK-2118 2700 μg IT Monotherapy | Arm 1 MK-2118 5400 μg IT Monotherapy | Arm 1 MK-2118 7700 μg IT Monotherapy | Arm 1 MK-2118 10000 μg IT Monotherapy | Arm 1 MK-2118 15000 μg IT Monotherapy | Arm 1 MK-2118 20000 μg IT Monotherapy | Arm 2 MK-2118 2700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 μg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Switch-over Arm 1 MK-2118 300 μg IT To Arm 2 900 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 2700 μg IT To Arm 2 2700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 5400 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 900 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 7700 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 15000 μg IT + Pembrolizumab 200 mg IV
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 14 | 12 | 4 | 8 | 12 | 7 | 5 | 3 | 3 | 3 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ng/mL | 2 (NA) — Method of dispersion could not be estimated due to n=1. | 2 (NA) — Method of dispersion could not be estimated due to n=1. | 3 (NA) — Method of dispersion could not be estimated due to n=1. | 3 (17) | 7 (70) | 6 (104) | 3 (90) | 8 (153) | 9 (105) | 7 (45) | 8 (99) | 6 (178) | 9 (127) | 10 (228) | 7 (142) | 7 (127) | 8 (168) | 5 (107) | 7 (44) | 44 (3435) | 11 (216) | 16 (212) | 36 (50) | 32 (64) |  |  |  |  |  |  |  |

5. Secondary Outcome: MK-2118 Maximum Plasma Concentration (Cmax)
Description: Cmax of MK-2118 was defined as the maximum concentration of MK-2118 observed in plasma. Blood samples were collected pre-dose and at specified timepoints post dose for estimation of MK-2118 Cmax. Per protocol, PK outcomes were not analyzed separately for the switch-over treatment arms.
Time Frame: as for outcome 4
Population: The subset of participants who complied with the protocol and had MK-2118 Cmax data available. Per protocol, PK outcomes were not analyzed separately for the switch-over treatment arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Arm 1 MK-2118 100 μg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 μg IT Monotherapy | Arm 1 MK-2118 900 μg IT Monotherapy | Arm 1 MK-2118 2700 μg IT Monotherapy | Arm 1 MK-2118 5400 μg IT Monotherapy | Arm 1 MK-2118 7700 μg IT Monotherapy | Arm 1 MK-2118 10000 μg IT Monotherapy | Arm 1 MK-2118 15000 μg IT Monotherapy | Arm 1 MK-2118 20000 μg IT Monotherapy | Arm 2 MK-2118 2700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 μg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Switch-over Arm 1 MK-2118 300 μg IT To Arm 2 900 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 2700 μg IT To Arm 2 2700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 5400 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 900 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 7700 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 15000 μg IT + Pembrolizumab 200 mg IV
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 14 | 12 | 4 | 8 | 12 | 7 | 5 | 3 | 3 | 3 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ng/mL | 6 (NA) — Method of dispersion could not be estimated due to n=1. | 75 (NA) — Method of dispersion could not be estimated due to n=1. | 94 (NA) — Method of dispersion could not be estimated due to n=1. | 259 (168) | 685 (41) | 1303 (57) | 1142 (91) | 2329 (84) | 3170 (47) | 442 (7) | 348 (568) | 1091 (99) | 1715 (60) | 1758 (242) | 790 (21) | 1530 (40) | 1630 (112) | 3032 (26) | 5441 (36) | 8407 (17) | 7168 (117) | 10637 (35) | 21763 (63) | 24117 (20) |  |  |  |  |  |  |  |

6. Secondary Outcome: MK-2118 Area Under the Concentration-time Curve From 0 to 24 Hours (AUC 0-24 Hours)
Description: AUC 0-24 hours of MK-2118 was defined as a measure of MK-2118 exposure that was calculated as the product of plasma drug concentration and time. Blood samples were collected pre-dose and at specified timepoints post dose for estimation of MK-2118 AUC0-24 hours. Per protocol, PK outcomes were not analyzed separately for the switch-over treatment arms.
Time Frame: as for outcome 4
Population: The subset of participants who complied with the protocol and had MK-2118 AUC0-24 hours data available. Per protocol, PK outcomes were not analyzed separately for the switch-over treatment arms.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*ng/mL
Arm/Group | Arm 1 MK-2118 100 μg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 μg IT Monotherapy | Arm 1 MK-2118 900 μg IT Monotherapy | Arm 1 MK-2118 2700 μg IT Monotherapy | Arm 1 MK-2118 5400 μg IT Monotherapy | Arm 1 MK-2118 7700 μg IT Monotherapy | Arm 1 MK-2118 10000 μg IT Monotherapy | Arm 1 MK-2118 15000 μg IT Monotherapy | Arm 1 MK-2118 20000 μg IT Monotherapy | Arm 2 MK-2118 2700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 μg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Switch-over Arm 1 MK-2118 300 μg IT To Arm 2 900 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 2700 μg IT To Arm 2 2700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 5400 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 900 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 7700 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 15000 μg IT + Pembrolizumab 200 mg IV
Number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 6 | 4 | 6 | 2 | 13 | 11 | 14 | 12 | 4 | 8 | 12 | 7 | 5 | 3 | 3 | 3 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
hour*ng/mL | 7 (NA) — Method of dispersion could not be estimated due to n=1. | 169 (NA) — Method of dispersion could not be estimated due to n=1. | 314 (NA) — Method of dispersion could not be estimated due to n=1. | 420 (181) | 1484 (36) | 2777 (59) | 2959 (92) | 4478 (34) | 6210 (47) | 944 (13) | 1217 (187) | 2300 (78) | 3219 (50) | 3993 (190) | 1630 (18) | 3272 (41) | 4518 (74) | 7736 (26) | 13866 (31) | 19257 (6) | 19946 (19) | 29638 (67) | 73573 (51) | 75171 (46) |  |  |  |  |  |  |  |

7. Secondary Outcome: Pembrolizumab Minimum Plasma Concentration (Cmin)
Description: Cmin of pembrolizumab was defined as the minimum concentration of pembrolizumab observed in plasma. Blood samples were to be collected at specified timepoints for estimation of pembrolizumab Cmin. Per protocol, analysis of pembrolizumab Cmin was not planned in Arm 1 (MK-2118 IT Monotherapy) or for the switch-over treatment arms. For Arm 2 (MK-2118 IT + Pembrolizumab combination) and Arm 4 (MK-2118 SC + Pembrolizumab combination), pembrolizumab Cmin data were not collected.
Time Frame: Predose on Day 1 of Cycles 1, 2, 3, 4, 5 and every 4 cycles thereafter (up to ~2 years) (Arm 2: length of Cycle= 3 weeks, Arm 4: length of Cycle 1= 2 weeks, length of Cycles 2 to 36= 3 weeks)
Population: The subset of participants who complied with the protocol and had pembrolizumab Cmin data available. Pembrolizumab Cmin analysis was not planned in Arm 1 (MK-2118 IT monotherapy) or for the switch-over treatment arms, per protocol. For Arm 2 (MK-2118 IT + Pembrolizumab combination) and Arm 4 (MK-2118 SC + Pembrolizumab combination), pembrolizumab Cmin data were not collected.
Arm/Group | Arm 1 MK-2118 100 μg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 μg IT Monotherapy | Arm 1 MK-2118 900 μg IT Monotherapy | Arm 1 MK-2118 2700 μg IT Monotherapy | Arm 1 MK-2118 5400 μg IT Monotherapy | Arm 1 MK-2118 7700 μg IT Monotherapy | Arm 1 MK-2118 10000 μg IT Monotherapy | Arm 1 MK-2118 15000 μg IT Monotherapy | Arm 1 MK-2118 20000 μg IT Monotherapy | Arm 2 MK-2118 2700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 μg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 μg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 μg SC + Pembrolizumab 200 mg IV Combination Therapy | Switch-over Arm 1 MK-2118 300 μg IT To Arm 2 900 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 2700 μg IT To Arm 2 2700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 5400 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 900 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 7700 μg IT To Arm 2 7700 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 10000 μg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 μg IT To Arm 2 15000 μg IT + Pembrolizumab 200 mg IV
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to ~65 months
Description: All-cause mortality (ACM): All allocated participants; AEs: All allocated participants who received ≥1 dose of study treatment. Per protocol disease progression of cancer was not considered an AE unless related to study drug. Thus, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression", "Disease progression" unrelated to study drug are excluded as AEs. Per protocol, ACM and AEs were analyzed separately for the switch-over treatment arms.
Arm/Group | Arm 1 MK-2118 100 µg Intra-tumoral (IT) Monotherapy | Arm 1 MK-2118 300 µg IT Monotherapy | Arm 1 MK-2118 900 µg IT Monotherapy | Arm 1 MK-2118 2700 µg IT Monotherapy | Arm 1 MK-2118 5400 µg IT Monotherapy | Arm 1 MK-2118 7700 µg IT Monotherapy | Arm 1 MK-2118 10000 µg IT Monotherapy | Arm 1 MK-2118 15000 µg IT Monotherapy | Arm 1 MK-2118 20000 µg IT Monotherapy | Arm 2 MK-2118 2700 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 5400 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 7700 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 10000 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 2 MK-2118 15000 µg IT + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 5000 µg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 10000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 15000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 20000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 30000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 45000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 60000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 90000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 120000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Arm 4: MK-2118 150000 µg SC + Pembrolizumab 200 mg IV Combination Therapy | Switch-over Arm 1 MK-2118 300 µg IT To Arm 2 900 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 2700 µg IT To Arm 2 2700 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 5400 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 900 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 7700 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV | Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 15000 µg IT + Pembrolizumab 200 mg IV
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 0/1 | 2/2 | 3/3 | 2/3 | 5/6 | 4/4 | 4/6 | 2/2 | 8/13 | 9/11 | 13/18 | 9/13 | 4/4 | 6/8 | 12/14 | 6/7 | 4/6 | 2/3 | 3/3 | 1/3 | 1/4 | 4/4 | 1/1 | 1/1 | 1/1 | 0/1 | 1/2 | 1/1 | 0/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 0/1 | 0/2 | 2/3 | 0/3 | 3/6 | 1/4 | 1/6 | 1/2 | 4/13 | 6/11 | 13/16 | 6/13 | 0/4 | 2/8 | 2/14 | 1/7 | 3/6 | 2/3 | 0/3 | 0/3 | 3/4 | 3/4 | 0/1 | 0/1 | 0/1 | 0/1 | 1/2 | 0/1 | 0/1 | 1/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 2/2 | 3/3 | 3/3 | 6/6 | 4/4 | 6/6 | 2/2 | 13/13 | 11/11 | 16/16 | 12/13 | 4/4 | 8/8 | 14/14 | 6/7 | 6/6 | 3/3 | 3/3 | 3/3 | 4/4 | 4/4 | 1/1 | 1/1 | 0/1 | 1/1 | 2/2 | 1/1 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 MK-2118 100 µg Intra-tumoral (IT) Monotherapy (N=1) | Arm 1 MK-2118 300 µg IT Monotherapy (N=1) | Arm 1 MK-2118 900 µg IT Monotherapy (N=1) | Arm 1 MK-2118 2700 µg IT Monotherapy (N=2) | Arm 1 MK-2118 5400 µg IT Monotherapy (N=3) | Arm 1 MK-2118 7700 µg IT Monotherapy (N=3) | Arm 1 MK-2118 10000 µg IT Monotherapy (N=6) | Arm 1 MK-2118 15000 µg IT Monotherapy (N=4) | Arm 1 MK-2118 20000 µg IT Monotherapy (N=6) | Arm 2 MK-2118 2700 µg IT + Pembrolizumab 200 mg IV Combination Therapy (N=2) | Arm 2 MK-2118 5400 µg IT + Pembrolizumab 200 mg IV Combination Therapy (N=13) | Arm 2 MK-2118 7700 µg IT + Pembrolizumab 200 mg IV Combination Therapy (N=11) | Arm 2 MK-2118 10000 µg IT + Pembrolizumab 200 mg IV Combination Therapy (N=16) | Arm 2 MK-2118 15000 µg IT + Pembrolizumab 200 mg IV Combination Therapy (N=13) | Arm 4: MK-2118 5000 µg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy (N=4) | Arm 4: MK-2118 10000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=8) | Arm 4: MK-2118 15000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=14) | Arm 4: MK-2118 20000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=7) | Arm 4: MK-2118 30000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=6) | Arm 4: MK-2118 45000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=3) | Arm 4: MK-2118 60000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=3) | Arm 4: MK-2118 90000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=3) | Arm 4: MK-2118 120000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=4) | Arm 4: MK-2118 150000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=4) | Switch-over Arm 1 MK-2118 300 µg IT To Arm 2 900 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 2700 µg IT To Arm 2 2700 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 5400 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 900 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 7700 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV (N=2) | Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 15000 µg IT + Pembrolizumab 200 mg IV (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Serositis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 MK-2118 100 µg Intra-tumoral (IT) Monotherapy (N=1) | Arm 1 MK-2118 300 µg IT Monotherapy (N=1) | Arm 1 MK-2118 900 µg IT Monotherapy (N=1) | Arm 1 MK-2118 2700 µg IT Monotherapy (N=2) | Arm 1 MK-2118 5400 µg IT Monotherapy (N=3) | Arm 1 MK-2118 7700 µg IT Monotherapy (N=3) | Arm 1 MK-2118 10000 µg IT Monotherapy (N=6) | Arm 1 MK-2118 15000 µg IT Monotherapy (N=4) | Arm 1 MK-2118 20000 µg IT Monotherapy (N=6) | Arm 2 MK-2118 2700 µg IT + Pembrolizumab 200 mg IV Combination Therapy (N=2) | Arm 2 MK-2118 5400 µg IT + Pembrolizumab 200 mg IV Combination Therapy (N=13) | Arm 2 MK-2118 7700 µg IT + Pembrolizumab 200 mg IV Combination Therapy (N=11) | Arm 2 MK-2118 10000 µg IT + Pembrolizumab 200 mg IV Combination Therapy (N=16) | Arm 2 MK-2118 15000 µg IT + Pembrolizumab 200 mg IV Combination Therapy (N=13) | Arm 4: MK-2118 5000 µg Subcutaneous (SC) + Pembrolizumab 200 mg IV Combination Therapy (N=4) | Arm 4: MK-2118 10000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=8) | Arm 4: MK-2118 15000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=14) | Arm 4: MK-2118 20000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=7) | Arm 4: MK-2118 30000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=6) | Arm 4: MK-2118 45000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=3) | Arm 4: MK-2118 60000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=3) | Arm 4: MK-2118 90000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=3) | Arm 4: MK-2118 120000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=4) | Arm 4: MK-2118 150000 µg SC + Pembrolizumab 200 mg IV Combination Therapy (N=4) | Switch-over Arm 1 MK-2118 300 µg IT To Arm 2 900 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 2700 µg IT To Arm 2 2700 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 5400 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 900 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 7700 µg IT To Arm 2 7700 µg IT + Pembrolizumab 200 mg IV (N=2) | Switch-over Arm 1 MK-2118 15000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 10000 µg IT + Pembrolizumab 200 mg IV (N=1) | Switch-over Arm 1 MK-2118 20000 µg IT To Arm 2 15000 µg IT + Pembrolizumab 200 mg IV (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 0 (0) | 3 (5) | 6 (7) | 0 (0) | 2 (2) | 0 (0) | 3 (6) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anisocoria (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 6 (7) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 6 (7) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (3) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 5 (6) | 3 (3) | 3 (3) | 0 (0) | 5 (5) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 3 (5) | 1 (1) | 0 (0) | 6 (13) | 3 (5) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 1 (1) | 2 (3) | 1 (1) | 5 (5) | 3 (3) | 4 (4) | 5 (5) | 2 (2) | 4 (4) | 5 (5) | 3 (3) | 3 (4) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 3 (3) | 4 (4) | 2 (5) | 0 (0) | 3 (6) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 1 (1) | 0 (0) | 3 (8) | 2 (4) | 4 (7) | 2 (2) | 6 (12) | 5 (6) | 6 (15) | 5 (9) | 1 (2) | 2 (4) | 3 (5) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 2 (5) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular device occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purulent discharge (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site irritation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 2 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour exudation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costovertebral angle tenderness (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/92/NCT03249792/Prot_SAP_000.pdf